CLINICAL TRIAL: NCT03608215
Title: Neuromodulation Effect of Transcranial Direct Current Stimulation in Severe Refractory Primary Dysmenorrhea: BDNF and MEG Study
Brief Title: Neuromodulatary Efficacy of Transcranial Direct Current Stimulation in Severe Refractory Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-01-005B
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Neuromodulation; Transcranial direct current stimulation; Neuroplasticity; Neuroimaging
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: active, sham
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): The anode sponge electrode will be placed on the scalp over the left primary motor cortex (M1) and the cathode sponge electrode will be positioned over the right supraorbital cortex (SO). Active stimulation consists of 2 mA current applied continuously for 20 minutes.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): The anode sponge electrode will be placed on the scalp over the left primary motor cortex (M1) and the cathode sponge electrode will be positioned over the right supraorbital cortex (SO). The 2 mA current will be applied for 30 seconds at the beginning of the session.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — The anode and cathode sponge electrode (51 cm2) will be placed over C3 and FP2 (10-20 system) respectively. 2 mA current will be applied continuously for 20 minutes.
  Arms: Active tDCS
Device: Sham tDCS — The anode and cathode sponge electrode (51 cm2) will be placed over C3 and FP2 (10-20 system) respectively. 2 mA current will be applied for 30 seconds at the beginning.
  Arms: Sham tDCS

SUMMARY:
Primary Dysmenorrhea (PDM), defined as menstrual pain without discernable organic causes, is inexorably common in adolescent women, about 40-90% of women may suffer from it, and 20% of them can be severe in the context of being refractory to medication, daily function impairment, and having pain of severe degree. Novel therapeutic method is in need for pain alleviation for this particular phenotype. It has been reported that PDM females may engage motor-cortex based descending pain modulation system in our resting-state functional Magnetic Resonance Imaging (rs-fMRI) and thermal pain-activation fMRI studies. Based on the reported analgesic efficacy of transcranial Direct Current Stimulation (tDCS) on the motor cortex for various experimental painful conditions and clinical pain disorders, it is plausible that tDCS can be effective for the severe and medication-refractory PDM patients. This study aim to investigate the analgesic efficacy of tDCS in severe PDMs and to elucidate the dynamic brain neuroplasticity in the context of experimental pain after tDCS intervention. Thirty severe PDMs will be recruited and randomly allocated to either real or sham group in a triple-blind manner. Experimental pain electrical stimulation will be performed before and after the tDCS intervention. The experimental pain-evoked magnetoencephamographic (MEG) data will be correlated with behavioral and psychological measurements. This is the first study in the literature investigating the tDCS efficacy for acute pain in severe PDM. The result can promise a new possibility for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 years old PDM patients
* Right-handedness
* A regular menstrual cycle: 27-32 days
* Cramping pain during the menstrual period in the last 6 months , VAS ≧ 7
* Abstinence for daily activities due to PDM
* Need analgesic or Physical therapy despite of no prominent effect

Exclusion Criteria:

* History of head injury
* Pathological pituitary gland disease
* Organic pelvic disease, psychiatric disorder
* Pregnancy, childbirth
* A metal or pacemaker implant.
* Take hormone agents within 6 months

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | change from baseline (1st menstrual phase, before tDCS) at one month (2nd menstrual phase, with tDCS), change from baseline (1st menstrual phase, before tDCS) at two months (3rd menstrual phase)
  pain scale; from 0 to 10; score 0: no pain, score 10: unbearable pain
Somatosensory evoked magnetic fields to experimental pain | change from baseline (before tDCS, before 2nd menstrual phase) at one week (after tDCS completion), change from baseline (before tDCS, before 2nd menstrual phase) at four weeks (before the 3rd menstrual phase)
  Somatosensory evoked magnetic fields (SEFs) is a well established magnetoencephalographic (MEG) cortical response evoked by electric stimulation. SEFs to experimental pain stimulation using electrical stimulator applied on the skin over the trajectory of median nerve will be used to evaluate pain-evoked cortical response.

SECONDARY OUTCOMES:
Quantitative sensory testing (QST) | change from baseline (before tDCS) at one week (after tDCS completion), change from baseline (before tDCS) at four weeks (before the 3rd menstrual phase), change from baseline (before tDCS) at five weeks (after the 3rd menstrual phase)
  To assess the threshold of thermal sensation (cold, cold-pain, heat, heat-pain; from 0 to 50 centigrade temperature), according to the established protocol of an ascending limit approach for heat pain and a descending limit approach for cold pain.
Spielberger State-Trait Anxiety Inventory (STAI) | change from baseline (before tDCS) at one week (after tDCS completion), change from baseline (before tDCS) at four weeks (before the 3rd menstrual phase), change from baseline (before tDCS) at five weeks (after the 3rd menstrual phase)
  To assess anxious symptoms; from 20 to 80; score 20: not anxious, score 80: extremely anxious
Beck Anxiety Inventory (BAI) | change from baseline (before tDCS) at one week (after tDCS completion), change from baseline (before tDCS) at four weeks (before the 3rd menstrual phase), change from baseline (before tDCS) at five weeks (after the 3rd menstrual phase)
  To assess anxious symptoms; from 0 to 63; score 0: not anxious, score 63: extremely anxious
Beck Depression Inventory (BDI) | change from baseline (before tDCS) at one week (after tDCS completion), change from baseline (before tDCS) at four weeks (before the 3rd menstrual phase), change from baseline (before tDCS) at five weeks (after the 3rd menstrual phase)
  To assess depressive symptoms; from 0 to 63; score 0: not depressed, score 63: extremely depressed
Pain Catastrophizing Scale (PCS) | change from baseline (before tDCS) at one week (after tDCS completion), change from baseline (before tDCS) at four weeks (before the 3rd menstrual phase), change from baseline (before tDCS) at five weeks (after the 3rd menstrual phase)
  To assess pain-maladaptive psychological status; from 0 to 52; score 0: not pain Catastrophizing , score 52: extremely pain Catastrophizing
Long-form McGill Pain Questionnaire (MPQ) | change from baseline (before tDCS) at one week (after tDCS completion), change from baseline (before tDCS) at four weeks (before the 3rd menstrual phase), change from baseline (before tDCS) at five weeks (after the 3rd menstrual phase)
  To assess pain status; from 0 to 78; score 0: not painful, score 78: extremely painful
Short-Form Health Survey (SF-36) | change from baseline (before tDCS) at one week (after tDCS completion), change from baseline (before tDCS) at five weeks (after the 3rd menstrual phase)
  To assess quality of life; he SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. From 0 to 100; score 0: equivalent to maximum disability, score 100: no disability.
Blood Hormones Measurement | change from baseline (before tDCS) at one week (after tDCS completion), change from baseline (before tDCS) at four weeks (before the 3rd menstrual phase)
  To assess testosterone, progesterone, estrogen
Genotyping | baseline
  To genotype the single nucleotide polymorphism genotyping (i.e., BDNF Val66Met polymorphism (rs6265), COMT Val158Met polymorphism (rs4680), OPRM1 (rs1799971), 5HTR2A (rs6313), SLC6A4 (rs25531)) from blood specimen
Efficacy of tDCS blinding | At 1 months after tDCS intervention
  To assure blinding efficacy; Patients do self-assessment about whether they receive real tDCS or sham tDCS. Assessment questionnaire:1 or 0. 1: real tDCS; 0: sham tDCS.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan